CLINICAL TRIAL: NCT02866916
Title: Phase I Study of SXL01 in Patients With Metastatic Castration-Resistant Prostate Cancer
Brief Title: Study of SXL01 in Patients With Metastatic Castration-Resistant Prostate Cancer (PROSTIRNA)
Acronym: PROSTIRNA
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study cancelled
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16GENH01
Record Dates: First submitted 2016-08-08; First posted 2016-08-15 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2016-11

CONDITIONS: Prostatic Cancer, Castration-Resistant
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation (Experimental): The standard method "3+3" will be used for dose escalation: the first 3 patients will be treated at level 1; consecutive cohorts of 3 to 6 patients will be treated with increasing doses of SXL01.
  Treatment will be administered until patient experiences unacceptable toxicity, PSA raising, progressive disease and/or treatment is discontinued at the discretion of the investigator or withdrawal of consent.
  Additional patients will be included at the Recommended Phase II Dose (RP2D) in the expansion phase.
  Interventions: Drug: SXL01

INTERVENTIONS:
Drug: SXL01 — Treatment will be administered continuously over 24h through the subcutaneous route.

SUMMARY:
This is a single site, open-label, non-randomized, dose escalation phase I study designed to evaluate the safety, the tolerability and the Recommended Phase II Dose (RP2D) of SXL01, a synthetic small interfering ribonucleic acid (RNA) targeting the androgen receptor messenger RNA (mRNA), in patients with metastatic castration-resistant prostate cancer.

A standard method "3+3" will be used for dose escalation. A maximum of 30 patients will complete the dose-escalation phase of the study; 12 additional patients will be included at the RP2D in the expansion phase.

ELIGIBILITY:
Inclusion Criteria:

1. Males age 18-80 years.
2. ECOG performance status 0 - 1.
3. Life expectancy of more than 3 months.
4. Histologically confirmed prostate adenocarcinoma without neuroendocrine differentiation or small cell feature.
5. Metastatic prostate cancer deemed to be unresponsive or refractory to hormone therapy.
6. Detectable metastases by bone scan, CT scan or MRI.
7. Surgically or medically castrated, with testosterone levels of < 50 ng/dL (< 2.0 nM). If the patient is being treated with LHRH agonists (patient who have not undergone orchiectomy), this therapy must have been initiated at least 4 weeks prior to Cycle 1 Day 1 and must be continued throughout the study.
8. Documented prostate cancer progression as assessed by the investigator with one of the following:

   8.1. PSA progression defined by a minimum of two raising PSA levels with an interval of >1 week between each determination. The PSA values at the screening visit must be ≥ 1 µg/l (1 ng/mL).

   8.2. Radiographic progression of soft tissue disease by modified RECIST criteria 1.1 or of bone metastasis with two or more documented new bone lesions on a bone scan with or without PSA progression.
9. Adequate hepatic, renal, and hematologic function: AST/ALT ≤ 2.5 X ULN; Normal bilirubin or ≤ 1.5 ULN in case of Gilbert's syndrome; Serum creatinine CL> 60 mL/min by the Cockcroft-Gault formula; Hemoglobin ≥ 10 g/dL; Absolute neutrophil count ≥ 1500/mm3, Platelet count ≥ 100,000/mm3.
10. Patients must have recovered from the toxic effects of prior therapy (except alopecia) to NCIC CTCAE version 4.03 grade ≤1 and to baseline laboratory values as defined in inclusion criteria 9.
11. If sexually active, willing to use barrier contraception during the treatment phase of the protocol.
12. Written informed consent and any locally required authorization (e.g., Social security for France (Health Insurance)) obtained from the patient prior to performing any protocol-related procedures, including screening evaluations.
13. Patient willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. BMI ≥ 30.
2. Evidence of brain metastasis.
3. Patient seropositive for HIV and/or hepatitis B antigen positive and/or Hepatitis C antibody.
4. Patient with history of autoimmune disease with the exception of vitiligo, psoriasis and controlled diabetes.
5. Active suspected or prior documented autoimmune disease (including inflammatory bowel disease, celiac disease, irritable bowel syndrome, Wegener's granulomatosis and Hashimoto's thyroiditis).
6. Patient with history of another malignancy, except for the following: skin cancers (melanoma excluded), previously treated cancer with no sign of disease for at least 3 years.
7. Patient with concurrent infection or concurrent chronic or acute illness such as pulmonary (asthma or COPD), cardiac (NYHA class III or IV) or hepatic disease, or other illness considered by the principal investigator to constitute an unwarranted high risk for investigational drug administration will be excluded.
8. Patient who has got a medical condition contraindicated for subcutaneous administration.
9. Chronic systemic corticosteroid use within 4 weeks of the first administration of SXL01 (more than 2 weeks for a dose > 0.5 mg/kg of prednisolone).
10. Treatment with any hormonal therapy or androgen antagonist, including flutamide, bicalutamide, nilutamide, ketoconazole, diethylstilbestrol, Abiraterone, or enzalutamide, within 4 weeks of the first administration with the exception of GnRH agonists.
11. Patients requiring a continuous curative anti-coagulant treatment.
12. Patients requiring a continuous bisphosphonate or denosumab treatment at inclusion. Note: the use of bisphosphonate and denosumab during the course of the study will be allowed.
13. Planned to initiate any other anti-tumor therapies during the study.
14. Radiation therapy or surgery within 4 weeks of the first administration of SXL01.
15. Mental impairment (psychiatric illness/social situations) that may compromise the ability of the patient to give informed consent and comply with the requirements of the study.
16. Patient who has forfeited his/her freedom by administrative or legal award or who is under guardianship.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of Dose Limiting Toxicities (DLT) during the first cycle of treatment with SXL01. | 25 months
Characteristics of Dose Limiting Toxicities (DLT) during the first cycle of treatment with SXL01. | 25 months
Incidence and severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 33 months
  Tolerability and safety will be assessed through recording of adverse events using National Cancer Institute Common Terminology Criteria for Adverse Event (NCI-CTCAE) toxicity classification, monitoring biological parameters and vital signs measurement.

SECONDARY OUTCOMES:
Preliminary efficacy endpoint : rate of patients presenting Prostate Specific Antigen (PSA) progression defined using Prostate Cancer Clinical Trial Working Group 3 (PCWG3) | 33 months
Preliminary efficacy endpoint : rate of patients presenting clinical or radiological progression using Response Evaluation Criteria in Solid Tumours (RECIST) V1.1 as defined by PCWG3. | 33 months
Pharmacokinetics - SXL01 plasma concentration | Cycle 1: pre-dose (T0) then 0.5, 3, 6, 24 hours post dose on day 1 ; T0 on days 4, 8, 15, 22. Subsequent cycles : before administration on day 1 (CXD1). The day of treatment discontinuation (CXDX) : 0.5, 1, 2, 24 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Pierre DELORD, MD, PhD, Principal Investigator — IUCT-O
Locations (1):
- Institut Claudius Regaud, Toulouse, France